CLINICAL TRIAL: NCT04631120
Title: Team-based Technology-enabled Integrated Patient/Caregiver-focused Dementia Study
Acronym: T2IP-DS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was never started and the PI is retiring.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Howard Kirshner, Vice Chair of Neurology, Professor and Director of Stroke Center, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 55555
Record Dates: First submitted 2020-11-10; First posted 2020-11-17 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): The proposed arm will involve an initial assessment using the Clinical Dementia Rating (CDR) Scale and Atherosclerotic Cardiovascular Disease (ASCVD) Risk Score for patients and Zarit Burden Interview (ZBI) for caregiver, followed by provision of standard educational material from the AA and Association for the Advancement of Retired Persons (AARP). Two phone sessions with a study nurse will occur post-enrollment in months 1 and 6 to discuss the educational material and perform a needs assessment; a summary of these and professional education on national evidence-based guidelines will be mailed to the patient's PCP of record. Education provided in this arm will be both patient- and caregiver-centered.
  Interventions: Other: Standard of Care
- Integrated Dementia Practice Unit Arm (Experimental): The integrated practice unit design is a coordinated, team-based, comprehensive, technology enabled, family focused care delivery design comprised of:
  * Dementia Central: Nurses, physicians, psychologists, social workers, and other relevant healthcare providers that will meet monthly to review participants progress and issues. Telehealth visits would facilitate home care.
  * Dementia Mobile: A nurse and lay health educator team will perform monthly visits, conduct assessments of subjects and provide education/coaching.
  * Dementia Link: Technologies that facilitate communication between Dementia Central and Dementia Mobile and foster proactive collaboration/coaching for study subjects include an mHealth software that allows for real time intervention/communication between professional teams and dyads, combined with management of dyads for multiple parameters like health metrics, behavioral measures and stress management and a portal tailored to specific clinical needs.
  Interventions: Other: Integrated Dementia Practice Unit Design

INTERVENTIONS:
Other: Integrated Dementia Practice Unit Design — * Dementia Central: monthly review of participant progress
  * Dementia Mobile: monthly nurse/lay health educator visits for assessments, education and coaching
  * Dementia Link: communication between Dementia Central and Dementia Mobile using the eTransX mHealth platform and HealthStream educational interface for care providers and the patient/caregiver dyad.
  Arms: Integrated Dementia Practice Unit Arm
Other: Standard of Care — Standard clinical practices of the physician and institution including an initial assessment, Zarit Burden Interview (ZBI) for caregiver, followed by provision of standard patient- and caregiver-centered educational material. Two phone sessions with a study nurse post-enrollment in months 1 and 6 to discuss the educational material and perform a needs assessment.
  Arms: Standard of Care

SUMMARY:
Dementia patients experience memory and other cognitive function deterioration leading to loss of independent function. Care required for dementia is multifactorial, spanning cognitive, behavioral, emotional, and physical symptoms, and complicates aspects of daily living. This places tremendous strain on caregivers who, in turn, experience their own increased physical and mental health needs. The current care model focuses primarily on patient pharmacological management but misses the mark on caregiver focus and collaboration. Building on systematic reviews and existing evidence gaps in information and support for patient/caregiver dyads, dealing with behavioral symptoms, referrals to available community resources, and multidisciplinary team care with improved coordination and communication17, the study investigators propose a patient- and caregiver-targeted Integrated Dementia Practice Unit (IDPU) model of care. IDPU integrates disconnected care under a centralized specialty team, providing monitoring, education, individualized support, and proactive, ongoing collaboration and coaching using technology and home/virtual visits for maximal impact. Days alive at home (DAAH) best captures quality of life (QOL) for the index dementia patient, from the perspective of both the healthcare system and the caregiver, and degree of support for the caregiver and is often an outcome in assessing health delivery. The study investigators hypothesize IDPU will increase DAAH and improve patient-level (behavioral; depressive symptoms; chronic disease management) and caregiver-level (strain, depressive symptoms, social support) outcomes relative to an Educational+ model, merging a standard care design with additional education support for patients/caregivers and their Primary Care Providers (PCP). This study seeks to (a) improve and establish IDPU feasibility of the in the feasibility phase, (b) determine if IDPU is more effective than Education+ in increasing DAAH and patient- and caregiver-level outcomes, and (c) determine if benefits of IDPU are more or less pronounced in vulnerable subgroups in the full-scale study.

ELIGIBILITY:
Inclusion Criteria include:

* Alzheimer's Disease or Vascular Dementia diagnosis provided by a study investigator
* 2 or 3 on the Clinical Dementia Rating Scale at time of enrollment
* Mini Mental Status Examination score of >10 or <25 administered at the time of enrollment
* Willingness and ability to provide patient or surrogate consent, and since caregiver cooperation will be an integral part of this study, an ability to provide caregiver consent to participate

Exclusion criteria include:

* Individuals with Mild Cognitive Impairment
* Institutionalized individuals (extended care facility, nursing home, group home, or similar institutional setting)
* Individuals who in the opinion of the investigator cannot be enrolled or followed due to geographic or other constraints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Days Alive and At Home | 12 months
  Our primary outcome is days alive at home (DAAH) for an index dementia patient within 1-year of enrollment (defined as days NOT in a hospital, extended care facility, in-patient rehabilitation, hospice, or respite care facility since enrollment).

SECONDARY OUTCOMES:
Number of Neurobehavioral Changes | 24 months
  Neurobehavioral changes measured by Neuro-Psychiatric Inventory, Cornell Scale for Depression in Dementia
Number of Health Resources Utilized | 24 months
  health resource contact-related outcomes (ER visits, office visits, urgent care or urgent office visits, respite care, hospitalizations for dementia-related illness)
Percent of Participants Achieving Chronic Disease Control Based on Risk Factor Averages | 24 months
  Chronic disease control at target for blood pressure, LDL-C (if hyperlipidemic), HbgA1c (if diabetic), exercise levels, BMI, diet
Perceived Social Support of Caregivers | 24 months
  Perceived social support using Multidimensional Scale of Perceived Social Support (Caregivers). 12-item measure of perceived adequacy of social support from three sources: family, friends, & significant other; using a 5-point Likert scale (0 = strongly disagree, 5 = strongly agree).
Assessment of Perceived Strain in Caregivers | 24 months
  Measurement of change in perceived strain in caregivers using Zarit Burden Interview. The ZBI uses a 4-point ordinal scale which describes the degree of burden being experienced from 0 = never to 4 = almost always. Maximum score is 88 and higher scores indicate more burden.
Assessment of Caregiver Stress | 24 months
  Measurement of change in caregiver stress using NPI Caregiver Distress Scale. Caregiver distress associated with the symptom is rated on an anchored 0- to 5-point scale identical to that used in the NPI. 12 The total NPI-Q distress score represents the sum of individual symptom scores and ranges from 0 to 60.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Kirshner, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No